CLINICAL TRIAL: NCT05270226
Title: Developing and Evaluating a Metacognitive ADHD Telehealth Intervention for Work-performance Enhancement (Work-MATE) Amongst Adults With ADHD
Brief Title: Metacognitive ADHD Telehealth Intervention for Work-performance Enhancement (Work-MATE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Rosenblum (Other)
Responsible Party: Sponsor-Investigator, Sara Rosenblum, Professor in the Department of Occupational Therapy, Faculty of Social Welfare, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Work-MATE
Record Dates: First submitted 2022-02-12; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: ADHD
Keywords: Work Performance; Occupational Performance; Executive Functions; Quality of Life; Organization in Time
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled and crossover trial to evaluate the evaluate the effect of the Work-MATE program on occupational performance at work of adults with ADHD.
  The first Intervention Group (A) received the Work-MATE intervention. After a crossover switching trial, the second Intervention Group (B) received the Work-MATE intervention in order. All evaluations were online, in similar environmental conditions.
  The Ethics Committee of the University of Haifa approved the study.
Who Masked: Participant, Care Provider
Masking Description: Participants were randomly assigned to Intervention Group A or B. Randomization sequence was created using permuted block design manually, with a 1:2 allocation, using block size of 6. The result of the randomization was blinded for participants and occupational therapists (OTs) who preformatted the intervention processes.
  Participants had not contact with other participants during all study phases. To address potential bias, all study assessments completed online, without involvement of the OTs who preformatted the intervention processes. The OTs and the participants were not exposed to baseline assessment scores or post-intervention scores of any study measure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): After being randomly allocated, group A participants had first evaluation (out of 3, pre-intervention) and immidiatlly recived Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE).
  Interventions: Behavioral: The Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE)
- Group B (Experimental): After being randomly allocated, group B participants had first evaluation (out of 4), then waiting-phase of 10-11 weeks, and after second evaluation (pre-intervention) start Work-MATE intervention process.
  Interventions: Behavioral: The Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE)

INTERVENTIONS:
Behavioral: The Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE) — The Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE) is an innovative program that aim to improve occupational performance at work of adults with ADHD, by enhancing their EF abilities, self-awareness, and personal strategy use.
  The Work-MATE is a short, synchronous and hybrid teleintervention program of eleven 1-hour weekly individual sessions. It offers a written standardized protocol, which include uniform structure of each intervention session and pool of therapy aids (for self-tailored matching by occupational therapists).

SUMMARY:
Adults with Attention-deficit hyperactivity disorder (ADHD) experience poor occupational performance at work compare to adults without ADHD, manifested at tendencies toward unemployment, job instability, work accidents, and sickness absences. This poor occupational performance at work may be partly caused by difficulties at executive functions (EF) abilities, and at the ability to set and attain goal directed work-activities at a satisfactory manner. Therefore, improvement at those abilities may followed by occupational performance at work enhancement of adults with ADHD. Such improvement may enhance adults with ADHD quality of life.

Despite the wide-ranging implications of poor occupational performance at work of adults with ADHD, treatments which focus at this component improvement among adults with ADHD are lack.

The Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE) is an innovative program that aim to improve occupational performance at work of adults with ADHD, by enhancing their EF abilities, self-awareness, and personal strategy use.

This program was established based on existing fundamental models and approach, (1) The World Health Organization's international classification of functioning, disability and health (ICF) (WHO, 2001), (2) Person-Environment-Occupation-Performance model (Baum, Christiansen, & Bass-Haugen, 2015) (3) The Dynamic Interactional Model of cognition (DIM; Toglia, 2018) and the Multicontex approach (Toglia, 2018) which based on the it, and (4) Telehealth as service-delivering model.

The Work-MATE aim to promote self-awareness and self-generation of personal strategies and increase efficiency strategy use across meaningful purposeful everyday work activities (i.e., goal directed work-activities). It is a short, synchronous and hybrid teleintervention program of eleven 1-hour weekly individual sessions, focused directly on occupational performance at work enhancement of adults with ADHD.

DETAILED DESCRIPTION:
Research Aim:

To develop and evaluate effectiveness of Metacognitive ADHD Telehealth intervention for Work-performance Enhancement (Work-MATE), of adults with ADHD.

Hypotheses:

The study sample (n=46) includes adults with ADHD, after confirmation of inclusion and exclusion criteria and symptoms consistency of ADHD. Participants enrolled randomly into two groups:

1. Group A (n=31)- received treatment immediately after the first assessment.
2. Group B (n =16)- was reassessed 10-11 weeks after the first assessment (the length of the treatment process), and then received treatment.

Both groups were reassessed at the end of the treatment (second assessment for group A and third assessment for group B). An additional assessment was performed three months after the end of treatment.

The hypotheses are presented in three stages:

Stage 1:

1. A comparison of the characteristics of study groups (A and B) participants as a preliminary stage to their unification as one group (n=46).

   Hypothesis 1: Differences will not be found in the demographic and occupational characteristics of participants when assessed using demographic and occupational questionnaires, and the ADHD characteristics using the Brown Attention-Deficit Disorder Scales (BADDS).
2. To examine the change in group B (n = 16) prior to treatment.

Hypothesis 2: Differences will not be found between assessment 1 and assessment 2 before the treatment in the following variables:

2. a. EF abilities- measured by Behavior Rating Inventory of Executive Function-Adult version (BRIEF-A) 2. b. occupational performance at work- evaluated by performance and satisfaction with performance scores as measured with the Canadian Occupational Performance Measure (COPM).

2. c. Quality of life- evaluated by Adult ADHD Quality of Life Questionnaire (AAQoL).

2. d. Organization in time ability- evaluated by Time Organization and Participation Scale (TOPS).

2. e. ADHD characteristics- evaluated by BADDS questionnaire.

Stage 2: Effectiveness of the Treatment

1. Examination of the effectiveness of the treatment process within both study groups (A and B) (n = 46), before and after treatment, and three months after its completion.

Hypothesis 3: Differences will be found in both study groups (research and comparison) before and after treatment, and after a follow-up assessment three months later, regarding:

3. a. EF abilities- measured by BRIEF-A. 3. b. occupational performance at work- evaluated by performance and satisfaction with performance scores as measured with the COPM.

3. c. Quality of life- evaluated by AAQoL. 3. d. Organization in time ability- evaluated by TOPS. 3. e. ADHD characteristics- evaluated by BADDS questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Participants worked at least 3 months at the same workplace.
2. Participants had formal medical diagnosis of ADHD.
3. Symptoms consistent with ADHD were confirmed either by the Adult ADHD Self-Report Scale (ASRS) version 1.1 (Kessler et al., 2005) final score or by medium-to-high probability of ADHD according to the BADDS (Brown, 2012).
4. Participants had at least one EF deficit according to the BRIEF-A (Roth et al., 2005).
5. Participants not receiving any functional additional treatment during the study period.
6. Participants read and write Hebrew fluently.

Exclusion Criteria:

People who self-reported comorbid mental health disorders, motor or neurological disabilities, chronic diseases, or significant injuries.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Canadian Occupational Performance Measure (COPM) at 3 and 6 months | Measure 1 (baseline; at third intervention meeting), measure 2 (after intervention completion; approximately 3 months from baseline), measure 3 (approximately 6 months from baseline)
  COPM used to evaluate self-perception of occupational performance at work. During semi-structured interview at the third session of intervention, the participant was asked to identify two meaningful activities for which he perceived the greatest performance problems during work, or activities that influence his occupational performance at work. Those two activities were set up as the two intervention goals. Participants rated each activity for performance from 1 (not able to do at all) to 10 (able to do extremely well) and similarly for satisfaction with performance. Significant improvement was considered as a change of at least two points between measures.
Change from Baseline Behavior Rating Inventory of Executive Function-Adult version (BRIEF-A) at 3 and 6 months | Measure 1 (baseline; 1 week before the beginning of the intervention), measure 2 (after the intervention completion; approximately 3 months from baseline), measure 3 (approximately 6 months from baseline)
  BRIEF-A measure EF abilities following the intervention. The score includes a global executive composite (GEC) index that represents the overall EF score, composed of a behavioral regulation index (BRI) score and a metacognition index (MI) score with nine nonoverlapping score scales. Scores of 65 or more for each index or scale indicate a clinical deficit.

SECONDARY OUTCOMES:
Change from Baseline Adult ADHD Quality of Life Questionnaire (AAQoL) at 3 and 6 months | Measure 1 (baseline; 1 week before the beginning of the intervention), measure 2 (after the intervention completion; approximately 3 months from baseline), measure 3 (approximately 6 months from baseline)
  AAQOL measures QoL of adults with ADHD, focusing on four domains: life productivity, psychological health, relationships, and life outlook. The AAQoL consists of 29 items rated on a 5-point scale for frequency of occurrence, which yields a total score and four subscale scores (reflecting the four domains). higher scores indicating better QoL.
Change from Baseline Time Organization and Participation Scale (TOPS) at 3 and 6 months | Measure 1 (baseline; 1 week before the beginning of the intervention), measure 2 (after the intervention completion; approximately 3 months from baseline), measure 3 (approximately 6 months from baseline)
  TOPS assesses the perceived ability of the individual to organize daily life tasks on time. Using this questionnaire three domains of organization on time had been evaluated: A, daily task performance at an appropriate pace; B, the individual's success in organizing a whole day or a certain period in a satisfactory manner; C, the frequency of emotional responses following disorganization in time. Because domain D items are used for clinical purposes, they not statistically analyzed in this study. In all domains, lower scores indicate higher risk of difficulties in organization and participation in time in daily tasks. Participants who had a mean final score less than 3.16 were considered to be at risk for difficulties in on-time organization of daily life tasks.
Change from Baseline Brown Attention-Deficit Disorder Scales (BADDS) at 3 and 6 months | Measure 1 (baseline; 1 week before the beginning of the intervention), measure 2 (after the intervention completion; approximately 3 months from baseline), measure 3 (approximately 6 months from baseline)
  BADDS measures a range of ADHD symptoms. The items are grouped into five clusters: organizing and activating to work, ssustaining attention and concentration, sustaining energy and effort, Managing Affective Interference, and utilizing working memory and accessing Recall. Clusters T scores greater than 65 is considered clinically significant

CONTACTS AND LOCATIONS:
Overall Officials: Sara Rosenblum, Prof., Study Director — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel